CLINICAL TRIAL: NCT01921647
Title: The Exploration for Pharmacodynamics and Pharmacokinetic Interaction Between YH4808, Amoxicillin and Clarithromycin in Healthy Subjects
Brief Title: The PK and PD Interaction Between YH4808, Amoxicillin and Clarithromycin in Healthy Subjects
Acronym: YH4808-108
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: YH4808-108
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: safety/tolerability and pharmacokinetics/pharmacodynamics
MeSH Terms: interventions — YH4808; Drugs, Investigational; Esomeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- YH4808, amoxicillin, clarithromycin (Experimental): single administration of YH4808 or amoxicillin or clarithromycin or YH4808 + amoxicillin + clarithromycin
  Interventions: Drug: YH4808; Drug: Amoxicillin; Drug: clarithromycin
- YH4808, amoxicillin and clarithromycin (Experimental): 7 days repeat administration of YH4808, amoxicillin and clarithromycin for H.pylori eradication
  Interventions: Drug: YH4808; Drug: Amoxicillin; Drug: clarithromycin
- YH4808 and amoxicillin (Experimental): 7 days repeat administration of YH4808 and amoxicillin for H.pylori eradication
  Interventions: Drug: YH4808; Drug: Amoxicillin
- nexium, amoxicillin and clarithromycin (Active Comparator): BID, 7 days repeat administration of nexium, amoxicillin and clarithromycin for H.pylori eradication
  Interventions: Drug: Nexium; Drug: Amoxicillin; Drug: clarithromycin

INTERVENTIONS:
Drug: YH4808
  Other Names: experimental drug
  Arms: YH4808 and amoxicillin; YH4808, amoxicillin and clarithromycin; YH4808, amoxicillin, clarithromycin
Drug: Nexium
  Other Names: active comparator
  Arms: nexium, amoxicillin and clarithromycin
Drug: Amoxicillin
  Other Names: experimental drug
Drug: clarithromycin
  Other Names: experimental drug
  Arms: YH4808, amoxicillin and clarithromycin; YH4808, amoxicillin, clarithromycin; nexium, amoxicillin and clarithromycin

SUMMARY:
The objective of this study is not only to explore pharmacokinetic interaction after single oral administration but also pharmacodynamics interaction after multiple oral administration of YH4808, amoxicillin and clarithromycin each separately versus coadministration of YH4808, amoxicillin and clarithromycin in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. healthy male age 20 to 55 over 55kg with Ideal body weight(BMI:18.5~25)
2. Subject who has no congenital, chronic disease and disease symptoms in medical examination result
3. Subject who is judged to be eligible by principal investigator or sub-investigator according to various reasons including their abnormal test results(clinical laboratory test, 12-lead GCG etc)

Exclusion Criteria:

1. Subject who is hypersensitive to components contained in YH4808 or this drug
2. Subject who has history or presence of clinically significant diseases in liver, kidney, gastrointestinal tract, nervous system, respiratory system, endocrine system, blood tumor, cardiovascular, urinary system, and mental disorder
3. Subject who has history of surgical operation or diseases related to gastrointestinal symptom (e.g. Crohn's disease, ulcer etc except appendectomy or simple for hernia)
4. Other exclusions apply

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Cmax, AUClast of YH4808, M3, amoxicillin, clarithromycin, 14-hydroxyclarithromycin | pre dose, 16 times after dosing

SECONDARY OUTCOMES:
Cmax, AUClast of M8, AUCinf, t1/2, Tmax of YH4808, M3, M8, amoxicillin, clarithromycin, 14-hydroxyclarithromycin | pre dose, 16 times after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Min soo Park, Ph.D, M.D., Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park H, Kim CO, Kim M, Lim Y, Lee WY, Yoon S, Park MS. Pharmacodynamic evaluation of YH4808 for Helicobacter pylori eradication in healthy subjects. Transl Clin Pharmacol. 2020 Sep;28(3):136-146. doi: 10.12793/tcp.2020.28.e16. Epub 2020 Sep 23. PMID 33062627
- [Derived] Lee WY, Oh E, Cui M, Kim CO, Lim Y, Kim H, Park H, Yoon S, Park MS, Hong T. Evaluation of pharmacokinetic interactions between amoxicillin, clarithromycin, and the potassium-competitive acid blocker YH4808 in healthy subjects. Transl Clin Pharmacol. 2020 Mar;28(1):55-65. doi: 10.12793/tcp.2020.28.e5. Epub 2020 Mar 31. PMID 32274381